CLINICAL TRIAL: NCT01853020
Title: Cannabinoids and Cerebellar-Motor Functioning
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1211011055
Record Dates: First submitted 2013-03-25; First posted 2013-05-14 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cannabis; Psychotic Disorders
Keywords: Cannabinoids; Eyeblink Conditioning; EBC
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THC (Active Comparator): Very low dose (0.0015 mg/kg = 0.21 mg in a 70 kg individual) THC, dissolved in alcohol. Administered intravenously over 10 minutes.
  Low dose (0.015 mg/kg = 1.05 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately ¼ of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  Medium dose (0.03 mg/kg = 2.1 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately ½ of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  Interventions: Drug: THC
- Placebo (Placebo Comparator): Control: small amount of alcohol intravenous (quarter teaspoon), with no THC over 10 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC — Very low dose (0.0015 mg/kg = 0.21 mg in a 70 kg individual) THC, dissolved in alcohol. Administered intravenously over 10 minutes.
  Low Dose (0.015 mg/kg = 1.05 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately ¼ of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  Medium dose (0.03 mg/kg = 2.1 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately ½ of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  Arms: THC
Drug: Placebo — Control: small amount of alcohol intravenous (quarter teaspoon), with no THC over 10 minutes.
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the dose-related effects of delta-9-tetrahydrocannabinol (∆9-THC) in healthy individuals on cerebellum-dependent motor functions.

DETAILED DESCRIPTION:
The overall aim of the current proposal is to investigate whether acute, IV ∆9-THC administration mediates cerebellar versus forebrain-dependent associative learning in humans as assessed with eyeblink conditioning (EBC). In addition, a battery of motor function tests will also be administered (the CANTAB motor screening test, Grooved Pegboard Motor Task, paced finger tapping).

ELIGIBILITY:
Inclusion Criteria:

* Must have used cannabis at least once in their lifetime
* No cannabis use in the past month
* Men and women aged 21 to 35 years (extremes included) on the day of the first dosing

Exclusion Criteria:

* Hearing deficits
* Psychiatric or mental disorders
* Hearing Deficits

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

PRIMARY OUTCOMES:
Cerebellum Dependent Associative Learning (% CRs) | Measured +15 minutes after infusion
  % conditioned responses (CRs) will be measured
Cerebellum Dependent Associative Learning (CR Latency) | Measured +15 minutes after infusion
  conditioned response (CR) Latency will be measured
Completion of the Grooved Pegboard Motor Task (Reaction Time/Accuracy) | Measured +45 minutes after infusion
  Total time taken to complete the grooved pegboard tasks will be the dependent measure.
CANTAB Motor Screening Test (Reaction Time) | Measured +45 minutes after infusion
  Using a touch screen, reaction time to touch a target will be the dependent measures.
CANTAB Motor Screening Test (Accuracy) | Measured +45 minutes after infusion
  Using a touch screen, accuracy to touch a target will be the dependent measures.
Paced Finger Tapping (Correct Responses) | Measured +45 minutes after infusion
  Using a button on a computer keyboard, correct responses will be measured.
Paced Finger Tapping (Reaction Time) | Measured +45 minutes after infusion
  Using a button on a computer keyboard, reaction time and tapping variability will be measured.

SECONDARY OUTCOMES:
THC intoxication, as measured by the Visual Analog Scale (Total Score) | Baseline; +45, +100, +240 minutes after infusion
  0 being none; 100 being completely

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States